CLINICAL TRIAL: NCT01185093
Title: St. Jude Cancer Education for Children Program: Evaluation at 4th-Grade Level
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SJCECP
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Cancer
Keywords: Cells; Prevention; Cancer education; Nutrition; Healthy living; Physical activity; Dangers of tobacco; Sun protection
MeSH Terms: conditions — Neoplasms; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Fourth grade students: Each participant will attend two presentations and six hands-on activities led by St. Jude faculty and research staff on topics within their expertise, such as cells and cancer, and healthy living. The pre-test will take place within 7±1 days before the program presentations and before students receive copies of the printed material. Two post-tests will take place. The first post-test will be administered within 7±1 days after the final scheduled program presentation and will be a measure of knowledge acquisition. The second post-test will take place 90±7 days post-intervention and will be a measure of knowledge retention.

SUMMARY:
The main objectives of the study is to

* Evaluate the knowledge acquisition and retention of 4th-grade students who participate in the St. Jude Cancer Education for Children Program
* To examine the relationship between outcome measures (knowledge acquisition and knowledge retention) with covariates of interest such as self-reported age and gender
* To compare the knowledge scores among schools and identify the schools that may show better improvement than others and factors associated with improvement

DETAILED DESCRIPTION:
The subjects in this research study will be current 4th-grade students at elementary schools in Memphis, Tennessee who choose to participate in the Program. These participants are not patients of St. Jude Children's Research Hospital. The Program will be implemented over a three-day period. Each student will attend two presentations and six hands-on activities led by St. Jude faculty and research staff on topics within their expertise, such as cells and cancer, and healthy living. Printed materials to be distributed as part of the St. Jude Cancer Education for Children Program have been developed by a multi-disciplinary team of St. Jude employees and local educators and reviewed by national experts for scientific accuracy and appropriate readability. Material includes three illustrated children's books, a laboratory manual, and activity sheets.

One pre- and two post-tests will be administered by designated school teachers. The tests consist of 10 multiple-choice questions per each of three modules(cells, cancer, and healthy living), validated by a group of experts for readability and content relevance. Knowledge acquisition will be assessed by taking the differences from first post-test to pre-test scores, obtained from 10 questions on each component of the intervention, and using one-sample signed rank test to evaluate the improvement in the knowledge scores. A similar analysis will be undertaken by taking the differences from the 2nd post-evaluation to the 1st post-evaluation for each participant to assess knowledge retention.

ELIGIBILITY:
Inclusion Criteria:

Study participants are not patients of St. Jude Children's Research Hospital.

* 4th-grade student
* Enrolled at a school participating in the St. Jude Cancer Education for Children Program

Exclusion Criteria:

* Student chooses not to participate in any or all of the activities and/or testing
* Request by a parent or guardian

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A convenience sample of schools that agree to participate in the St. Jude Cancer Education for Children Program. 2-3 public schools and 2-3 private schools will be selected in order to achieve a fair representation of the Mid-South area. Based on average class sizes, this study expects to enroll at least 200 public school students and about 100 private school students.
Sampling Method: Non-Probability Sample
Enrollment: 481 (Actual)
Dates: Start 2010-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
This study will measure knowledge acquisition and retention of 4th grade students. | 1 year
  Knowledge acquisition will be assessed by taking the differences from first post-test to pre-test scores, obtained from 10 questions on each component of the intervention. A similar analysis will be undertaken by taking the differences from the 2nd post-evaluation to the 1st post-evaluation for each participant to assess knowledge retention.

SECONDARY OUTCOMES:
This study will measure age and gender | 1 year
  The study will examine the relationship between outcome measures(knowledge acquisition and knowledge retention) with covariates of interest such as self-reported age and gender.
This study will measure the knowledge scores among schools | 1 year
  To compare the knowledge scores among schools and identify the schools that may show better improvement than others and factors associated with improvement

CONTACTS AND LOCATIONS:
Overall Officials: Yuri Quintana, Ph.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St . Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org